CLINICAL TRIAL: NCT02727205
Title: A Multiple Site Study to Evaluate the Irritation and Sensitization Potential of Repeat Applications of Rotigotine Transdermal System, 1 mg/24 hr Versus Neupro (Rotigotine Transdermal System), 1 mg/24 hr in Healthy Volunteers
Brief Title: Irritation and Sensitization Potential of Repeat Applications of Rotigotine Patch
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inflamax Research Incorporated (Industry)
Responsible Party: Principal Investigator, Piyush Patel, MD, Medical Director, Inflamax Research Incorporated
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AC13GP01
Record Dates: First submitted 2016-02-25; First posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Bioequivalence - Irritation and Sensitization Potential of Transdermal Patch
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): One-half (½) of the test patch and one-half (½) of the reference patch (Rotigotine Transdermal System) was applied daily to the same site for each product over a 21 day period followed by a 14 day rest phase and a 48 hour challenge phase.
  Interventions: Drug: Rotigotine Transdermal System

INTERVENTIONS:
Drug: Rotigotine Transdermal System
  Other Names: Neupro

SUMMARY:
STUDY TITLE:

A Multiple Site Study to Evaluate the Irritation and Sensitization Potential of Repeat Applications of Rotigotine Transdermal System, 1 mg/24 hr Versus Neupro (Rotigotine Transdermal System), 1 mg/24 hr in Healthy Volunteers

TEST DRUG / INVESTIGATIONAL PRODUCT:

Rotigotine Transdermal System, 1 mg/24 hr

INDICATION STUDIED:

Bioequivalence - Irritation and Sensitization

STUDY DESIGN:

* Multiple-site, randomized, multiple-application, evaluator-blinded, controlled study
* One-half (½) of the test patch and one-half (½) of the reference patch was applied daily to the same site for each product over a 21 day period followed by a rest phase and a challenge phase

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and non-pregnant female volunteers. All subjects were healthy, non-smoking male and female (nonpregnant) volunteers between the ages of 18 and 65, who were demonstrated to be generally healthy by screening medical and medication history, physical examinations, vital signs, 12-lead electrocardiogram (ECG), and FSH levels (if applicable).

Exclusion Criteria:

1. Reported receiving any investigational drug within 30 days prior to Day 1 patch application.
2. Reported a clinically significant illness during the 28 days prior to Day 1 patch application (as determined by the Investigator[s]).
3. Reported a history of allergic response(s) to rotigotine or related drugs.
4. Reported a history of sulfite sensitivity.
5. Demonstrated a clinically relevant finding, as determined by the clinical Investigator(s), on the screening ECG, such as a second- or third-degree atrioventricular block or complete bundle branch block, or arrhythmias.
6. Reported a history of asthma, orthostatic hypotension, dizziness, syncope, or dyskinesia. At the discretion of the Principal Investigator, subjects with a history of asthma or mild asthma not requiring regular treatment could have been included.
7. Systolic blood pressure < 100 or >145 mmHg or diastolic blood pressure < 60 or > 95 mmHg at screening measured in supine position after 5 minutes rest; heart rate < 50 or > 100 at screening.
8. Reported a history of narrow angle glaucoma.
9. Reported the use of monoamine oxidase (MAO) inhibitors, reserpine, methyldopa, antipsychotics, neuroleptics, benzodiazepines, antidepressants, clozapine, olanzapine, quetiapine, metoclopramide, or risperidone within 3 months of enrollment.
10. Reported a history of somnolence and/or of falling asleep without warning.
11. Reported a history of significant dermatologic diseases or conditions such as atopy, or psoriasis.
12. Reported a history of medical conditions known to alter skin appearance or physiologic response (eg diabetes, porphyria).
13. Reported a history of significant dermatologic cancers (eg melanoma, squamous cell carcinoma). Basal cell carcinomas that were superficial and did not involve the investigative sites were acceptable.
14. Reported a history of conditions that would significantly influence the immune response (e.g. primary or acquired immunodeficiencies such as HIV positive or AIDS, or generalized drug reaction, neoplasms such as lymphoma or leukemia, moderate or severe rheumatoid arthritis or active systemic lupus erythematosus).
15. Demonstrated an obvious difference in skin color amongst application sites, presence of a skin condition, excessive hair (subjects that agreed to have their hair clipped short [not shaved] prior to patch application were eligible), scar tissue, recent sunburn, tattoo, open sore, body piercing, or branding at the intended sites of application that would interfere with placement of study articles, skin assessment or reactions to drug.
16. Reported the use of any immunosuppressive drugs, including systemic and topical corticosteroids and retinoids within 28 days prior to Day 1 patch application.
17. Reported the use of any medications or treatments that would significantly influence or exaggerate responses to the patches or that would alter inflammatory or immune responses to the patches within 21 days prior to Day 1 patch application (e.g. cyclosporine, tacrolimus, systemic or topical corticosteroids, cytotoxic drugs, immune globulin, Bacillus Calmette-Guerin [BCG], monoclonal antibodies, radiation therapy).
18. Reported the use of any anti-inflammatory medication, including ibuprofen and Celebrex, within 72 hours of Day 1 patch application, with the exception of steroid nose drops and/or eye drops.
19. Reported the use of antihistamines or topical drugs at the patch site within 72 hours of Day 1 patch application.
20. Reported a history of anaphylactic reaction to drugs. At the discretion of the Investigator, subjects with seasonal allergic rhinitis with sensitivity to environmental allergens could have been included.
21. Reported a history of sensitivity or allergy to adhesive bandages, tapes, or transdermal systems.
22. Reported a significant history of allergy to soaps, lotions, emollients, ointments, creams, cosmetics, adhesives, or latex.
23. Reported a history of drug or alcohol addiction or abuse within the past year.
24. Was pregnant, lactating, breastfeeding, or intended to become pregnant over the course of the study (females only).
25. Demonstrated a positive pregnancy screen (females only). Subjects with a positive result at screening were to be excluded from the study. Subjects with a positive result during the study were to be withdrawn.
26. Reported smoking or using tobacco products or was currently using nicotine products (patches, gums, etc.). Ninety (90) days abstinence was required.
27. Reported a plan to undergo magnetic resonance imaging or cardioversion procedures during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Irritation | 21 days (Induction Phase)
  The primary endpoint of cumulative irritation was the measurement of the combined "Dermal response" and "Other Effect" total irritation scores recorded during the 21 day continuous application period (i.e. the total irritation score for a specific subject was the sum of the irritation scores recorded on Days 2 through 22 for each patch type). Because the cumulative irritation scores did not display a normal distribution, the primary analysis was a comparison of the overall median of the observed total irritation score of the Test patch against the Reference patch. The Per Protocol Population for Irritation (PPPI) was used for the primary analysis
Sensitization | 48 and 72 hour post removal of patch after the challenge phase.
  The primary analysis of sensitization used the Per Protocol Population for Sensitization (PPPS) and compared the number and percentage (%) of reactions indicating potential sensitization (irritation score greater than or equal to 2 at 48 or 72 hours post-removal, along with the Investigator's assessment) observed with each patch type

SECONDARY OUTCOMES:
Adhesion | 21 days (Induction Phase) and 1 day Sensitization Phase
  Adhesion scores

CONTACTS AND LOCATIONS:
Locations (2):
- Clinical Pharmacology of Miami, Inc., Miami, Florida, United States
- Inflamax Research Inc., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No